CLINICAL TRIAL: NCT05462314
Title: An Evaluation of the Intestinal Microbiome, Oral Microbiome, and Whole Blood Transcriptome Analyses in Gastrointestinal Malignancies
Brief Title: Intestinal Microbiome, Oral Microbiome, and Whole Blood Transcriptome Analyses in Gastrointestinal Malignancies
Status: Completed | Type: Observational
Sponsor: Viome (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: V130
Record Dates: First submitted 2022-07-07; First posted 2022-07-18 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Cancer; Pancreatic Cancer; Esophageal Cancer; Gastric Cancer; Rectal Cancer; Liver Cancer; Biliary Cancer
Keywords: gastrointestinal cancer; GI cancer; metastatic cancer; microbiome; pancreas; esophagus; rectum; liver
MeSH Terms: conditions — Gastrointestinal Neoplasms; Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Rectal Neoplasms; Liver Neoplasms; Biliary Tract Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Gastrointestinal Malignancies (pancreatic, colorectal, gastroesophageal, and hepatobiliary): Individuals with a gastrointestinal malignancy including pancreatic, colorectal, gastroesophageal, or hepatobiliary malignancies.

SUMMARY:
The primary objective of this prospective observational study is to characterize the gut and oral microbiome as well as the whole blood transcriptome in gastrointestinal cancer patients and correlate these findings with cancer type, treatment efficacy and toxicity. Participants will be recruited from existing clinical sites only, no additional clinical sites are needed.

DETAILED DESCRIPTION:
The primary objective of this prospective observational study is to characterize the gut and oral microbiome as well as the whole blood transcriptome in gastrointestinal cancer patients and correlate these findings with cancer type, treatment efficacy and toxicity.

This study will provide biospecimens from a diverse range of gastrointestinal cancer patients to allow preliminary characterization of the diversity and composition of the GIM microbiome and pilot analysis of changes in the microbiome as a function of both treatment and disease progression.

This is a prospective cohort study will characterize and evaluate the microbiome of GIM patients, with various histologies. The investigators plan to enroll 200 patients with a diagnosis of gastrointestinal cancer including pancreatic, esophageal, gastric, colon, rectal, liver and biliary cancers with (i) newly diagnosed recurrent or metastatic disease initiating therapy or (ii) with progressive disease on second or later line therapies, or (iii) with locally advanced, inoperable disease receiving palliative therapy. Stool, blood and saliva samples will be collected at baseline, early in treatment (3-6 weeks), and then at 3 month intervals until progression or intolerable toxicity or up to 36 months.

The results of this study are expected to provide the basis for larger, more focused studies of the microbiome in distinct GIMs and relationship to specific treatment efficacy and toxicity. Ultimately, this classification of the gastrointestinal cancer microbiome may lead to novel risk stratification paradigms, novel treatments and maintenance strategies. Furthermore, this study may lead to improved diagnostics, companion diagnostics, and nutritional interventions for cancer prevention and therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of gastrointestinal malignancy including pancreatic, esophageal, gastric, colon, rectal, hepatocellular, or biliary carcinoma.
* Subjects must have a) newly diagnosed recurrent or metastatic disease b) progressive disease on second or later line therapies, or c) locally advanced inoperable disease receiving palliative therapy.
* Age > 18 years.
* Ability to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Subjects with gastrointestinal malignancy already receiving treatment including chemotherapy, immunotherapy, radiation therapy or investigational agents for treatment of a) newly diagnosed recurrent or metastatic disease b) progressive disease on second or later line therapies, or c) locally advanced disease.
* Subjects with gastrointestinal malignancy who will not be receiving cancer directed therapy including chemotherapy, immunotherapy, radiation therapy or investigational agents.
* Subjects with active infectious gastroenteritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will accrue subjects being treated for gastrointestinal malignancies (pancreatic, colorectal, gastroesophageal, and hepatobiliary) at MSSM who are receiving chemotherapy and/or immunotherapy. Male and female subjects, between 18 and 100 years of age, who agree to donate blood, saliva, and stool specimens taken for research purposes in the outpatient setting are eligible. The elderly will be included since many gastrointestinal malignancies affect the elderly. Subjects with known active systemic infections will be excluded due to potential laboratory contamination of other resources.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Characterization of the microbiome in Gastrointestinal Malignancy | 3 years
  Determining the number of species present in the sample.
Levels of gene expression of the identified species in Gastrointestinal Malignancy | 3 years
  Determining the levels of gene expression in the species found.

SECONDARY OUTCOMES:
Relationship between treatment efficacy and microbiome diversity | 3 years
  Determination of the relationship between treatment efficacy and microbiome diversity, composition and function. Changes (increase or decrease) to the number of species and changes (increase or decrease) to their genetic expression as a result of their treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Guruduth Banavar, Principal Investigator — Viome
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No